CLINICAL TRIAL: NCT03019029
Title: Diagnostic Utility of F-18 Florbetapir PET/MR in Peripheral Nerve Amyloidosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Stephen M. Broski, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 16-006798
Record Dates: First submitted 2017-01-03; First posted 2017-01-12 (Estimated); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Amyloidosis
Keywords: Peripheral Nerve Amyloidosis
MeSH Terms: conditions — Amyloidosis

STUDY DESIGN:
Intervention Model Description: Participants with biopsy proven peripheral nerve amyloidosis will undergo an F-18 Florbetapir PET/MR scan
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Peripheral nerve amyloidosis (Experimental): Patients with pathologically-confirmed peripheral nerve amyloidosis will undergo 18-F Florbetapir PET/MR scan on a GE SIGNA PET/MR scanner.
  Interventions: Other: 18-F Florbetapir PET/MR scan

INTERVENTIONS:
Other: 18-F Florbetapir PET/MR scan — 18-F Florbetapir PET/MR scan, PET/MR on a GE SIGNA PET/MR scanner

SUMMARY:
The primary aim of this study will be to examine the diagnostic utility of 18-F Florbetapir PET/MR (Positron Emission Tomography/Magnetic Resonance) in imaging patients with pathologically-confirmed systemic amyloidosis involving the peripheral nerves and compare these results to non-amyloid diseased controls.

DETAILED DESCRIPTION:
Patients with pathologically proven amyloidosis involving the peripheral nervous system will undergo 18-F Florbetapir PET/MR on a GE (General Electric Healthcare) SIGNA PET/MR scanner. A control arm comprised of patients with pathologically-confirmed non-amyloid causes of peripheral neuropathy will also undergo 18-F Florbetapir PET/MR scanning. all images will be reviewed for peripheral nerve uptake.

ELIGIBILITY:
Inclusion Criteria:

* Adults: 18-100
* Pathologically-confirmed peripheral nerve amyloidosis or pathologically-confirmed non-amyloid causes of peripheral neuropathy

Exclusion Criteria:

* Metallic devices that are not MR safe (cardiac pacers, stents, aneurysm coils, etc.)
* Claustrophobia
* BMI over 38

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2017-03-13 (Actual); Primary Completion 2022-03-22 (Actual); Study Completion 2022-03-22 (Actual)

PRIMARY OUTCOMES:
Locations of peripheral nerve 18-F Florbetapir uptake | 50-120 minutes post injection
  Standardized uptake value (SUV)
Pattern of F-18 Florbetapir uptake (Heterogeneous vs. Homogeneous, focal vs. diffuse) | 50-120 minutes post injection
  Heterogeneous vs. Homogeneous, focal vs. diffuse. This is a categorical variable. There is not a quantitative or semi-quantitative scale that is appropriate.

SECONDARY OUTCOMES:
T1 and T2 characteristics (Hypointense, isointense or hyperintense relative to skeletal muscle) | 50-120 minutes post injection
  Hypointense, isointense or hyperintense relative to skeletal muscle. This is a categorical variable. There is not a quantitative or semi-quantitative scale that is appropriate.
Morphologic changes | 50-120 minutes post injection
  Presence or absence of neural enlargement
Pattern of contrast enhancement (Solid, heterogeneous or peripheral enhancement) | 50-120 minutes post injection
  Solid, heterogeneous or peripheral enhancement. This is a categorical variable. There is not a quantitative or semi-quantitative scale that is appropriate.
Additional sites of 18-F Florbetapir uptake | 50-120 minutes post injection
  i.e. cardiac myocardium, skeletal muscle, bone marrow

CONTACTS AND LOCATIONS:
Overall Officials: Stephen M. Broski, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials